CLINICAL TRIAL: NCT07143214
Title: Wise Eating: A Guided Digital DBT-Based Intervention for Binge Eating-A Randomized Controlled Trial
Brief Title: Wise Eating: A Guided Digital DBT-Based Intervention for Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-YJ09
Record Dates: First submitted 2025-08-11; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Bulimia Nervosa; Binge Eating Behaviour; Anorexia Nervosa; Eating Disorders
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder; Anorexia Nervosa; Feeding and Eating Disorders | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital DBT group (Experimental)
  Interventions: Behavioral: online dialectical behavior therapy
- Waitlist control (Placebo Comparator): waitlist patient is provided with psychoeducation
  Interventions: Behavioral: Waitlist and psychoeducation

INTERVENTIONS:
Behavioral: online dialectical behavior therapy — Enrolled participants will be provided with credentials to access the mobile application for a 28-day therapist-supported DBT self-help intervention. Participants are required to engage with the application at least once daily throughout the 4-week intervention period, with each session requiring approximately 30 minutes of engagement. The application delivers automated daily reminders at user-configurable timepoints. Additionally, participants receive asynchronous text-based guidance via WeChat during the treatment phase, wherein therapists provide support, feedback, and clinical direction during predetermined response windows. Each participant's cumulative weekly guidance duration is capped at 15 minutes.
  The application's therapeutic framework integrates core components from The Dialectical Behavior Therapy Skills for Emotional Eating and standardized DBT treatment manuals, structured across four evidence-based modules: (1) Mindfulness, (2) Distress Tolerance, (3) Interpersonal Eff
  Arms: Digital DBT group
Behavioral: Waitlist and psychoeducation — The active control group serves as a rigorous placebo comparator condition. Participants allocated to this arm will receive daily psychoeducational communications regarding binge-eating pathology, encompassing epidemiological data, biopsychosocial determinants, clinical manifestations, and therapeutic approaches. Crucially, all disseminated content remains devoid of Dialectical Behavior Therapy (DBT)-related components or skill-building elements.
  Arms: Waitlist control

SUMMARY:
Bulimia Nervosa (BN), characterized by binge eating and purging behaviors, constitutes a chronic psychiatric disorder predominantly affecting young females, characterized by high prevalence and relapse rates. Its core features include recurrent binge-eating episodes accompanied by compensatory behaviors such as self-induced vomiting and laxative misuse, resulting in significant impairment to patients' physiological, psychological, and social functioning. Recent epidemiological trends in China indicate a rising BN incidence, with suspected prevalence rates reaching 4.7%-17% among secondary and tertiary education cohorts.

Nevertheless, current treatment modalities present substantial concerns. Despite established evidence-based clinical practice guidelines, merely 25% of affected individuals receive appropriate intervention. Multiple systemic barriers impede care access, including: (1) scarcity of adequately trained clinicians; (2) patient-endorsed stigma and apprehension regarding eating disorders (EDs); (3) geographical constraints; (4) financial burdens associated with in-person therapy; and (5) insufficient treatment-seeking motivation.

The proliferation of mobile technologies has positioned mHealth as a viable solution to expand patient coverage. This modality offers self-diagnostic, monitoring, and therapeutic opportunities for populations with limited access to traditional care, while simultaneously mitigating treatment-related stigmatization. Consequently, this project investigates the efficacy of a Dialectical Behavior Therapy (DBT)-based self-help system for binge-eating behaviors. Employing a randomized controlled trial (RCT) design, BN patients will be allocated to intervention and control groups. Comparative analysis of clinical psychological metrics will be conducted at baseline, 2-week, 4-week, and 8-week intervals post-intervention, with feasibility assessed through structured interviews. This research aims to establish an effective, low-cost remote self-help intervention to enhance treatment accessibility and therapeutic outcomes for BN patients.

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfill all following conditions:

(i) Aged ≥18 years; (ii) Proficient in operating WeChat-enabled smartphones; (iii) Exhibit binge-eating behaviors: ≥4 binge-eating episodes within the preceding 28-day period; (iv) If receiving psychotropic medication: stable dosing regimen maintained for ≥1 month prior to enrollment, with no planned dosage adjustments during the trial period; concurrent psychotherapy is exclusionary; (v) Absence of structured nutritional therapy or formal psychological interventions within 30 days preceding enrollment; (vi) Demonstrated comprehension of the study protocol and provision of written informed consent.

Exclusion Criteria:

(i) Severe anxiety or depressive symptom. (ii) Investigator-determined contraindications to trial participation based on clinical assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
BES, Binge Eating Scale | Baseline, treatment period (4 weeks) post-treatment (4 weeks past day 1.), 1 month follow up after treatment, 3 months follow up after treatment

SECONDARY OUTCOMES:
DERS, Difficulties in Emotion Regulation Scale | Baseline, treatment period (4 weeks) post-treatment (4 weeks past day 1.), 1 month follow up after treatment, 3 months follow up after treatment
PHQ, Patient Health Questionnaire | Baseline, treatment period (4 weeks) post-treatment (4 weeks past day 1.), 1 month follow up after treatment, 3 months follow up after treatment
GAD, Generalized Anxiety Disorder 7-item scale | Baseline, treatment period (4 weeks) post-treatment (4 weeks past day 1.), 1 month follow up after treatment, 3 months follow up after treatment
BIS, Barratt Impulsiveness Scale | Baseline, treatment period (4 weeks) post-treatment (4 weeks past day 1.), 1 month follow up after treatment, 3 months follow up after treatment
EDE-Q, Eating Disorder Examination Questionnaire | Baseline, treatment period (4 weeks) post-treatment (4 weeks past day 1.), 1 month follow up after treatment, 3 months follow up after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Likely share upon reasonable request